CLINICAL TRIAL: NCT01596959
Title: The Contact-CTI Study - Does Assessment of Tissue Contact During Ablation of Atrial Flutter Improve Outcomes?
Brief Title: The Contact-CTI Study: Use of Tissue Contact Data to Guide Atrial Flutter Ablation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 79426/244082/1/568; 11/SC/0394 (Other: NRES Oxford C south central)
Record Dates: First submitted 2012-05-09; First posted 2012-05-11 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2012-05

CONDITIONS: Atrial Flutter
Keywords: atrial flutter; ablation; irrigation; contact; ECI
MeSH Terms: conditions — Atrial Flutter | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ECI CONTACT-ACTIVE (Active Comparator): Irrigated Radiofrequency ablation performed using the ECI contact data
  Interventions: Procedure: Radiofrequency ablation utilising the ECI contact software
- ECI CONTACT-INACTIVE (Placebo Comparator): irrigated RF ablation performed to the right atrium without the use of ECI contact data
  Interventions: Procedure: Radiofrequency ablation without the use of ECI contact data

INTERVENTIONS:
Procedure: Radiofrequency ablation utilising the ECI contact software — irrigated radiofrequency ablation to the right atrium using the ECI contact data
  Other Names: Ensite Contact; Electrical Coupling Index
  Arms: ECI CONTACT-ACTIVE
Procedure: Radiofrequency ablation without the use of ECI contact data — irrigated RF ablation without the use of ECI contact data
  Arms: ECI CONTACT-INACTIVE

SUMMARY:
This study will be a single blind prospective randomised control trial in patients undergoing ablation for the treatment of typical atrial flutter, with the aim of investigating the benefit of a new impedance-based computer software application which measures tissue contact between the ablation catheter and the inside of the heart.

The investigators hope to demonstrate that the use of this tissue contact information reduces ablation time, Xray time, and procedure time required to complete the procedure successfully. Study participants will be randomly assigned to undergo their procedure with or without this contact data displayed for the doctor performing the ablation to see. The acute procedural endpoint of ablation is successful conduction block across the cavotricuspid isthmus of the right atrium. If the outcome of this study is positive, it will have a significant beneficial impact on this procedure, reducing procedure length, patient discomfort, and potentially reducing risk for the patient, recurrent arrythmia symptoms, and the need for repeat procedures later on.

DETAILED DESCRIPTION:
Patients in this study will be de novo cases of atrial flutter ablation, and they will be randomised to ablation using tissue contact data provided by the St. Jude medical ECI technology (active arm), or standard ablation as per physician practice, without the use of contact data to guide ablation (control arm). The endpoint measures will include RF ablation time, procedure time, time to achieving cavotricuspid isthmus block, the need for "touch up" ablation to achieve conduction block, the recurrence rate of isthmus conduction on isuprel infusion at 20 minutes post-isolation, and clinical recurrence of atrial flutter post-operatively.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is undergoing de novo cavotricuspid isthmus ablation.
2. Participant is willing and able to give informed consent for participation in the study.
3. Male or Female, aged 18 years or over

Exclusion Criteria:

(1) Previous percutaneous or open surgical procedure involving the right atrium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2012-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the mean ablation time required to achieve the acute procedural endpoint of cavotricuspid isthmus conduction block | immediate (intra-procedural)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Betts, MbChB, MD, Study Director — Oxford University Hospitals NHS Trust
Locations (1):
- John Radcliffe Hospital, Headington, Oxfordshire, United Kingdom